CLINICAL TRIAL: NCT05717881
Title: Impact of Poplar Propolis on Insulin Homeostasis and Pancreatic Cell Function in Insulin Resistant Subjects
Brief Title: Impact of Poplar Propolis on Metabolic Disturbances of Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aix Marseille Université (Other)
Collaborators: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Principal Investigator, Jean-Francois Landrier, Principal Investigator, Aix Marseille Université
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 1
Record Dates: First submitted 2023-01-27; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Insulin Resistance
Keywords: Propolis
MeSH Terms: conditions — Insulin Resistance | interventions — Propolis

STUDY DESIGN:
Intervention Model Description: The present trial was a randomized, double-bind, controlled, crossover, dietary intervention study. During this trial, two types of supplementations were randomly administered during two treatment periods (propolis and placebo), using a random number table. The placebo served as the reference group for comparison. Participants and caregivers were blinded to the type of treatment consumed.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propolis (Experimental): Propolis supplements were packaged in marine capsules and consisted of poplar propolis powder (propolis concentrate, carob powder, magnesium stearate and silicon dioxide), concentrated to 30% total polyphenols.
  Each supplementation period lasted 3 months, with a 2-week wash-out period, to allow total excretion of polyphenols by the body and do not interfere with the new supplementation phase.
  The subjects in this study were submitted to five visits, allowing the tracking of biological parameters (clinical examination, fasting blood samples, HGPO) during the study. During the supplementation phases, follow-up by telephone call was performed.
  Interventions: Dietary Supplement: Propolis
- Placebo (Placebo Comparator): Placebo powder capsules (maltodextrin, fatty acids, magnesium salts and silicon dioxide) are presented in the same packaging to have an identical appearance and taste. Patients in the propolis group were dosed with propolis to reach 6 mg total polyphenols/kg body weight, based on the results of a previous preclinical study in mice.
  Each supplementation period lasted 3 months, with a 2-week wash-out period, to allow total excretion of polyphenols by the body and do not interfere with the new supplementation phase.
  The subjects in this study were submitted to five visits, allowing the tracking of biological parameters (clinical examination, fasting blood samples, HGPO) during the study. During the supplementation phases, follow-up by telephone call was performed.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Propolis — Propolis supplements were packaged in marine capsules and consisted of poplar propolis powder (propolis concentrate, carob powder, magnesium stearate and silicon dioxide), concentrated to 30% total polyphenols.
  Each supplementation period lasted 3 months, with a 2-week wash-out period, to allow total excretion of polyphenols by the body and do not interfere with the new supplementation phase.
  The subjects in this study were submitted to five visits, allowing the tracking of biological parameters (clinical examination, fasting blood samples, HGPO) during the study. During the supplementation phases, follow-up by telephone call was performed.
  Arms: Propolis
Dietary Supplement: Placebo — Placebo powder capsules (maltodextrin, fatty acids, magnesium salts and silicon dioxide) are presented in the same packaging to have an identical appearance and taste. Patients in the propolis group were dosed with propolis to reach 6 mg total polyphenols/kg body weight, based on the results of a previous preclinical study in mice.
  Each supplementation period lasted 3 months, with a 2-week wash-out period, to allow total excretion of polyphenols by the body and do not interfere with the new supplementation phase.
  The subjects in this study were submitted to five visits, allowing the tracking of biological parameters (clinical examination, fasting blood samples, HGPO) during the study. During the supplementation phases, follow-up by telephone call was performed.
  Arms: Placebo

SUMMARY:
Propolis, a natural resinous mixture rich in polyphenols, produced by bees from a variety of plant sources, has shown significant therapeutic effects and may prevent the development of certain chronic diseases. Current evidence supports the beneficial effect of these bioactive phytochemicals on the management of type 2 diabetes mellitus (T2DM) and other chronic diseases. The objective of this study is to evaluate the effect of poplar propolis extract powder (PPEP) on glucose homeostasis and other clinical parameters in insulin-resistant patients (diagnosed by HOMA-IR index > 1.85 for men and > 2.07 for women).

DETAILED DESCRIPTION:
Backgroud: Propolis, a natural resinous mixture rich in polyphenols, produced by bees from a variety of plant sources, has shown significant therapeutic effects and may prevent the development of certain chronic diseases. Current evidence supports the beneficial effect of these bioactive phytochemicals on the management of type 2 diabetes mellitus (T2DM) and other chronic diseases. The objective of this study is to evaluate the effect of poplar propolis extract powder (PPEP) on glucose homeostasis and other clinical parameters in insulin-resistant patients (diagnosed by HOMA-IR index > 1.85 for men and > 2.07 for women).

Methods: The trial was a randomized, controlled, crossover, intervention study. Insulin-resistant patients (n=9) (8 women, 1 man), with a mean ± SD age 49 ± 7, were subjected to two periods of supplementation (propolis and placebo) for 3-months, separated by a 2-week washout period. The quantity of propolis administered was determined individually to reach 6 mg of polyphenols/kg. Fasting blood test and oral glucose tolerance test (OGTT) were performed before and after each treatment.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥ 30 kg/m2
* Insulin resistance defined as a HOMA-IR index > 1.85 for men and > 2.07 for women

Exclusion Criteria:

* Presence of diabetes
* Recent weight change (≥ 5% in the last 3 months)
* Documented allergy to bee products and/or fish products
* Positive serology for human immunodeficiency virus or hepatitis
* High blood pressure
* Elevated transaminases (AST > 40 IU/L ; ALT > 45 IU/L)
* Low creatine clearance (estimated glomerular filtration rate < 90 ml/min)
* Interfering treatment (cholesterol-lowering treatment, intestinal absorption modulating treatment, absorption modulating treatment and/or insulin sensitivity)
* Gastrointestinal tract surgery
* Pregnancy and / or lactation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Change in the Matsuda-DeFronzo Insulin Sensitivity Index (ISI-M) | 3 months
  The primary outcome was change in the Matsuda-DeFronzo Insulin Sensitivity Index (ISI-M) at the end of supplementation. The ISI-M is calculated by the following formula: 10,000 / square root [(Glu0 × Ins0) × (Glumean OGTT × Insmean OGTT)], where Glux and Insx represent plasma glucose (mg/dL) and insulin values (UI/L), respectively, at time x min during. The ISI-M index, proposed by Matsuda and Defronzo, makes it possible to estimate insulin sensitivity derived from the OGTT

SECONDARY OUTCOMES:
Change in glucose homeostasis | 3 months
  Glycaemia at T0, T30, T60, T90 and T120 (mmol/L) mesured after after an oral glucose tolerance test (OGTT).
Change in insulin homeostasis | 3 months
  Insulinemia at T0, T30, T60, T90 and T120 (mUI/L) mesured after after an oral glucose tolerance test (OGTT).
Change in triglyceride levels | 3 months
  Enzymatic assay by spectrophotometry of triglycerides (mmol/L).
Change in cholesterol levels | 3 months
  Enzymatic assay by spectrophotometry of cholesterol (mmol/L).
Change in high density lipoprotein (HDL) cholesterol levels | 3 months
  Enzymatic assay by spectrophotometry of HDL cholesterol (mmol/L).
Change in low density lipoprotein (LDL) cholesterol levels | 3 months
  Friedewald formula : LDL=cholesterol-HDL-(triglyceride/2,2) expressed in mmol/L.
Change in glycated hemoglobin A1c (HbA1c) levels | 3 months
  HbA1c mass spectrometry assay (%).
Change in weight | 3 months
  Weight measurement by scale (kg).
Change in body mass index (BMI) | 3 months
  BMI calculated by weight (kg) / size (m) squared.
Change in body fat rate | 3 months
  Fat mass rate estimated by impedancemetry (DEXA) (%).
Change in body lean rate | 3 months
  Lean mass rate estimated by impedancemetry (DEXA) (%).
Change in C-reactive protein | 3 months
  Enzymatic determination of CRP (mg/L).
Change in transaminases levels | 3 months
  Enzymatic determination of alanine aminotransferase (ALAT) and aspartate aminotransférase (ASAT) (UI/L).
Change in gamma glutamyl transferases (GGT) | 3 months
  Enzymatic determination of gamma glutamyl transferases (GGT) (UI/L).
Change in 8-iso-prostaglandin F2α levels | 3 months
  Enzymatic determination of 8-iso-prostaglandin F2α (8-iso-PGF 2α) (pg/mL).
Change in creatinine levels | 3 months
  Enzymatic determination of creatinine (mg/L).
Change in creatinine clearance | 3 months
  Estimation of creatinine clearance (mL/min) by formula : 1,23 (for men) or 1,04 (for women) x weight (kg) x (140 - age)/creatinine (mg/L).
Change in leptin levels | 3 months
  Enzymatic determination of leptin (pg/mL).
Change in adiponectin levels | 3 months
  Enzymatic determination of adiponectin (ng/mL).

CONTACTS AND LOCATIONS:
Overall Officials: Jean Francois Landrier, PhD, Principal Investigator — Aix Marseille Université
Locations (1):
- CIC La conception, Marseille, France